CLINICAL TRIAL: NCT06873217
Title: Acupuncture for Dizziness and Vertigo in Emergency Department: a Single-center, Self-control, Observational Clinical Study During 2019-2023
Brief Title: Acupuncture for Dizziness and Vertigo in Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Yu-Chen Lee, Director of Department of Acupuncture, China Medical University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH113-REC1-066
Record Dates: First submitted 2025-03-02; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Dizziness and Vertigo
MeSH Terms: conditions — Dizziness; Vertigo | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Acupuncture + Western medical care Group (Experimental): Once a patient with Vertigo and Dizziness came to the emergency department, emergency physicians ask if they were willing to accept acupuncture intervention in addition to the routine western medical care.
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Once a patient with Vertigo and Dizziness came to the emergency department, emergency physicians ask if they were willing to accept acupuncture intervention in addition to the routine western medical care.

SUMMARY:
This study was conducted at China Medical University Hospital, Taiwan, between January 2019 and December 2023, with 345 patients diagnosed with dizziness and vertigo (ICD-10 codes R42 and H81). Patients received acupuncture in addition to standard Western medical care. The Visual Analogue Scale (VAS) was used to assess symptom severity before and after the acupuncture intervention. Secondary analyses explored the influence of ICD-10 classification, gender, and seasonality on treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

Patients who were diagnosed as ICD number R42 and H81

Exclusion Criteria:

Patients who were not suitable to accept acupuncture or refused to accept acupuncture

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale (VAS) change | 30 minutes
  The primary outcome in this study was the difference of Visual Analogue Scale (VAS) before and after intervention, aiming to assess if patient's condition got better after acupuncture.
  VAS is one of the pain rating scales, with the minimum value 0 and the maximum value 10, used for the first time in 1921 by Hayes and Patterson. From the patient's perspective, this spectrum appears continuous; their pain does not take discrete jumps, as a categorization of none, mild, moderate and severe would suggest. It was to capture this idea of an underlying continuum that the VAS was devised.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University, Taichung, Taiwan